CLINICAL TRIAL: NCT00496821
Title: A Study to Investigate the Safety and Efficacy of Intranasal ALN-RSV01 Administered to Adult Volunteers Experimentally Inoculated With Respiratory Syncytial Virus
Brief Title: Intranasal ALN-RSV01 Administered to Adult Volunteers Experimentally Inoculated With Respiratory Syncytial Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALN-RSV01-105
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ALN-RSV01

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of intranasal ALN-RSV01 versus placebo, administered once daily for 5 days to a healthy male volunteers experimentally inoculated with RSV

ELIGIBILITY:
Inclusion Criteria:

* Availability for the required study period (including the inpatient phase, ability to comply with study requirements and attend follow-up study visits
* Able to provide written consent for participation after reading the Consent Form and after having adequate opportunity to discuss the study with an investigator or qualified deputy.
* Good general health status as determined by a screening evaluation no greater than 120 days but not less than 14 days prior to enrollment and admission to the research unit
* Low titers of RSV neutralizing antibody measured during screening.

Exclusion Criteria:

* Significant acute or chronic, uncontrolled medical illness
* Presence of household member or close contact to someone who:

  * Is less than three(3) years of age
  * Has a known immunodeficiency
  * Is receiving immunosuppressant drugs
  * Is undergoing or soon to undergo cancer chemotherapy within 28 days of enrollment
  * Has diagnosed emphysema, chronic obstructive pulmonary disease(COPD), or severe lung disease
  * Is elderly and residing in a nursing home, or
  * Has received an organ transplant
* Females are not eligible for this study
* Evidence of or history of drug or alcohol abuse (within the past 6 months) or positive urine drug or alcohol screen

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2007-07; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of intranasal ALN-RSV01 versus placebo, administered in a multiple-dose schedule (once daily for 5 days) to healthy adult volunteers experimentally inoculated with respiratory syncytial virus | 28 days

SECONDARY OUTCOMES:
Determining the impact of ALN-RSV01 on symptoms of RSV infection, RSV infection rate based upon measures of viral load, and understanding the potential antiviral activity of ALN-RSV01 | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Akshay Vaishnaw, MD PhD, Study Director — Alnylam Pharmaceuticals
Locations (1):
- Alnylam Pharmaceuticals, Cambridge, Massachusetts, United States